CLINICAL TRIAL: NCT00649207
Title: A Phase 1 Study Evaluating the Safety, Tolerability and Pharmacokinetics of ABT-888 in Combination With Whole Brain Radiation Therapy in Subjects With Brain Metastases
Brief Title: A Phase I Study of ABT-888 in Combination With Conventional Whole Brain Radiation Therapy (WBRT) in Cancer Patients With Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-128
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2013-05

CONDITIONS: Brain Diseases; Brain Neoplasms; Central Nervous System Diseases; Neoplasm Metastasis; Nervous System Neoplasms
Keywords: WBRT; Brain Metastases; Radiation; ABT-888; PARP
MeSH Terms: conditions — Brain Diseases; Brain Neoplasms; Central Nervous System Diseases; Neoplasm Metastasis; Nervous System Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is an open label study; therefore, there are no numbered/labeled study arms.
  This is a dose escalation study, ABT-888 dose will be escalated in conjunction with two schedules of whole brain radiation therapy (WBRT). Subjects may be treated WBRT for 3 weeks (15 days) or 2 weeks (10 days).
  Interventions: Drug: ABT-888; Radiation: Whole Brain Radiation Therapy

INTERVENTIONS:
Drug: ABT-888 — Oral Capsules
  Other Names: veliparib
Radiation: Whole Brain Radiation Therapy — 15 fractions of 2.5 Gy over 3 weeks to a total dose of 37.5 GY or 10 fractions of 3.0 Gy over 2 weeks to a total dose of 30 Gy
  Other Names: WBRT

SUMMARY:
This Phase I clinical trial is studying the side effects and best dose of ABT-888 when given together with Whole Brain Radiation Therapy (WBRT) in treating patients with brain metastases.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, dose-escalation study evaluating the safety, tolerability and pharmacokinetics of the PARP inhibitor ABT-888 in combination with conventional whole brain radiation therapy (WBRT) in the treatment of subjects with solid tumors metastatic to the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age is greater than or equal to 18 years.
* Histologically or cytologically confirmed non-CNS primary solid malignancy.
* Pathologically or radiographically confirmed metastatic disease in the brain. Subjects with non-measurable lesions, including leptomeningeal carcinomatosis, are eligible.
* WBRT is clinically indicated, with the exception of prophylactic treatment.
* Karnofsky Performance Status (KPS) greater than or equal to a score of 70.
* Adequate hematology, renal and hepatic function.
* Both men and women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 2 months following completion of protocol therapy.

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
  * A vasectomized partner * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
  * Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* Subject is capable of understanding and complying with parameters as outlined in the protocol.
* Subject or the subject's legally acceptable representative has voluntarily signed and dated the informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Brain metastases secondary to germ cell tumor or lymphoma malignancy.
* Primary central nervous system (CNS) neoplasm.
* Prior or concurrent administration of the following therapies or treatments:

  * Prior treatment with WBRT
  * SRS performed less than 14 days prior to WBRT D1, or is scheduled to occur within 30 days of the last WBRT session
  * Last dose of chemotherapy, immunotherapy, biologic therapy, or investigational therapy was less than 14 days prior to WBRT D1. Bisphosphonates, hormone modification therapy, and trastuzumab are permitted without restriction
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or prior anti-cancer treatment.
* Known seizure disorder (status epileptics) that is uncontrolled, or seizures occurring greater than or equal to 3 times a week over the past month.
* If female, subject is pregnant or breast-feeding.
* Clinically significant and uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal, hematologic or neurological/psychiatric disease or disorder, including but not limited to:

  * Active uncontrolled infection
  * Symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
  * Any other illness condition(s) that could exacerbate potential toxicities, confound safety assessments, require excluded therapy for management, or limit compliance with study requirements
* Unable to swallow and retain oral medications.
* Known contraindication to enhanced MRI and CT, including but not limited to:

  * Presence of metal objects within the body such as a cardiac pacemaker, implanted cardiac defibrillator, brain aneurysm clips, cochlear implant, ocular foreign body, or shrapnel
  * History of immediate or delayed hypersensitivity reaction or other contraindication to contrast agents including but not limited to gadolinium and iodine
* Previous enrollment in this study or another study involving the investigation of ABT-888, with the exception of receiving a single dose of study drug.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-888 and/or WBRT.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of ABT-888 in combination with whole brain radiation therapy | ABT-888 will be dose escalated until the largest dose is reached that is felt to be safe based on safety information from all subjects.

SECONDARY OUTCOMES:
Safety Assessment Physical and Neurological Exam | be performed at all study visits, final and follow-up visit
Safety Assessment Mini-Mental State Examination | be performed at all study visits, final and follow-up visit
Safety Assessment Laboratory testing | be performed at all study visits, final and follow-up visit
  Chemistry and Hematology labs will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Shepherd L Stacie, MD, Study Director — AbbVie
Locations (9):
- United States (7):
  - Site Reference ID/Investigator# 8334, Atlanta, Georgia
  - Site Reference ID/Investigator# 52462, Chicago, Illinois
  - Site Reference ID/Investigator# 24483, Kansas City, Kansas
  - Site Reference ID/Investigator# 7180, Baltimore, Maryland
  - Site Reference ID/Investigator# 19021, Detroit, Michigan
  - Site Reference ID/Investigator# 6344, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6653, Madison, Wisconsin
- Site Reference ID/Investigator# 18542, Toronto, Canada
- Site Reference ID/Investigator# 46322, Ponce, Puerto Rico

REFERENCES:
- [Result] Mehta MP, Wang D, Wang F, Kleinberg L, Brade A, Robins HI, Turaka A, Leahy T, Medina D, Xiong H, Mostafa NM, Dunbar M, Zhu M, Qian J, Holen K, Giranda V, Curran WJ. Veliparib in combination with whole brain radiation therapy in patients with brain metastases: results of a phase 1 study. J Neurooncol. 2015 Apr;122(2):409-17. doi: 10.1007/s11060-015-1733-1. Epub 2015 Feb 15. PMID 25682091